CLINICAL TRIAL: NCT04113902
Title: The Effects of Health Education About Human Papilloma Virus and Cervical Cancer Prevention on Knowledge, Attitudes, Beliefs and Behaviors of Adolescent Girls and Their Mothers: A Prospective Randomized Controlled Study
Brief Title: The Effects of Health Education About Human Papilloma Virus and Cervical Cancer Prevention on Knowledge, Attitudes, Beliefs and Behaviors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Serpil Ozdemir, PhD, RN, Assistant Professor, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018/15- 18/331
Record Dates: First submitted 2019-08-02; First posted 2019-10-03 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2018-12

CONDITIONS: Health Education
Keywords: Human Papilloma Virus vaccine; Health education; Nursing; Adolescent Health
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Health education is given intervention group and 12 weeks follow up.
  Interventions: Behavioral: Health Education
- control group (No Intervention): Control group takes standard health care and 12 weeks follow up.

INTERVENTIONS:
Behavioral: Health Education — the adolescent girls and their mothers who participated in the intervention group were given health education twice in the first interview and in the fifth week. Follow-up continued for 12 weeks. The adolescent girls and their mothers in the control group received routine clinical practice. The effects of health education were evaluated with Human Papilloma Virus Knowledge Scale and Health Belief Model Scale for Human Papilloma Virus and its Vaccination.
  Arms: intervention group

SUMMARY:
Aim: To determine the effects of health education about Human Papilloma Virus infection and cervical cancer prevention on knowledge, attitudes, beliefs and behaviors of adolescent girls and their mothers.

Background: To combat with cervical cancer, it is urgent that prevention Human Papilloma Virus related disease all around the world.

Design: A randomized trial with a control group (n=108) and an intervention group (n=108).

Methods: The study was applied between January to June 2019 in the two different adolescent outpatient clinics in Turkey. The outpatient clinics were randomly assigned as intervention and control groups by numbering and opaque and sealed envelopes. Based on the intention-to-treat principle, all participants were analyzed according to the group they were assigned to, regardless of whether they received the intervention or not. In addition to the routine clinical practice, the adolescent girls and their mothers who participated in the intervention group were given health education twice in the first interview and in the fifth week. Follow-up continued for 12 weeks. The adolescent girls and their mothers in the control group received routine clinical practice. The effects of health education were evaluated with Human Papilloma Virus Knowledge Scale and Health Belief Model Scale for Human Papilloma Virus and its Vaccination.

Impact: Human Papilloma Virus vaccine, which has an important place in primary protection from cervical cancer, is expected to provide effective results by facilitating access to vaccine accompanied with health education.

ELIGIBILITY:
Inclusion Criteria:

To be a girl between the ages of 9 and 18, to be a mother of a girl between the ages of 9 and 18, to be fluent in Turkish, to be literate

Exclusion Criteria:

to be male, to have previously received Human Papilloma Virus vaccination, to have hearing, speech impairment and mental disorder, not to follow the study regularly, to use medication due to psychotic treatments, to be an adolescent with sexual experience

Min Age: 9 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 216 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Health Belief Model Scale for Human Papilloma Virus and Vaccine | three months
  In the four-point Likert scale, each item is scored between "none = 1" and "too much = 4.. The lowest score is 14 and the highest score is 56.
Human Papilloma Virus Knowledge Scale | three months
  True 1 "points are given to the correct answers given by the participants to each item, and" 0 "points are given to wrong and undecided' 'answers with incorrect answers. The lowest score that can be obtained from the scale is "0" and the highest is "10".

SECONDARY OUTCOMES:
Human Papilloma Virus Knowledge Scale | three months
  rue 1 "points are given to the correct answers given by the participants to each item, and" 0 "points are given to wrong and undecided' 'answers with incorrect answers. The lowest score that can be obtained from the scale is "0" and the highest is "10".
Health Belief Model Scale for Human Papilloma Virus and Vaccine | three months
  In the four-point Likert scale, each item is scored between "none = 1" and "too much = 4.. The lowest score is 14 and the highest score is 56.

CONTACTS AND LOCATIONS:
Locations (1):
- Serpil Özdemir, Ankara, Turkey (Türkiye)